CLINICAL TRIAL: NCT04301232
Title: Fast-Track Eligibility and Hospital Discharge for Outpatient Lumbar Discectomy: A Prospective Observational Study
Brief Title: Fast-Track Eligibility and Hospital Discharge for Outpatient Lumbar Discectomy
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mehmet Burak Eşkin, Assistant professor, Gulhane School of Medicine
Other Study IDs: 18/148
Record Dates: First submitted 2020-03-04; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Lumbar Disc Disease; Post-Op Complication
Keywords: PACU-bypass; hospital discharge; lumbar discectomy
MeSH Terms: conditions — Intervertebral disc disease; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fast-Track Group: After extubation, patients were evaluated using modified Aldrete Scoring System (mASS) , White's Fast- Track Scoring System (WFTSS) and SPEEDS criteria during 15 minutes with 3 min intervals. Patients who fulfilled criteria of all scoring systems were defined as eligible for PACU by-pass (fast-tracking) and transferred into phase II recovery area in the ward without observation in PACU (Group FT = Fast Track;)
  Interventions: Other: Modified Aldrete Scoring System (mASS); Other: White's Fast-Track Scoring System (WFTSS); Other: SPEEDS criteria
- PACU Group: After extubation, patients were evaluated using modified Aldrete Scoring System (mASS) , White's Fast- Track Scoring System (WFTSS) and SPEEDS criteria during 15 minutes with 3 min intervals. Ineligible patients were taken into PACU where their treatments were continued until discharge criteria were achieved (Group PACU)
  Interventions: Other: Modified Aldrete Scoring System (mASS); Other: White's Fast-Track Scoring System (WFTSS); Other: SPEEDS criteria

INTERVENTIONS:
Other: Modified Aldrete Scoring System (mASS) — Activity( Moves all extremities, Moves two extremities, Unable to move extremities), Respiration( Breathes deeply, coughs freely, Dyspneic, shallow or limited breathing, Apneic), Circulation (blood pressure) ( 20 mm Hg > preanesthetic level, 20 - 50 mm Hg > preanesthetic level, 50 mm Hg > preanesthetic level), Consciousness (Fully awake, Arousable on calling, Not responding), Oxygen saturation( SpO2 > 92% on room air, Supplemental O2 required to maintain SpO2 > 90%,SpO2 < 90% with O2 supplementation), scoring is done as 2,1,0, respectively. A score of 9 or more would be required for a patient after general anesthesia for discharge
Other: White's Fast-Track Scoring System (WFTSS) — Physical activity (Able to move all extremities on command, ,Some weakness in movement of extremities, Unable to voluntarily move extremities),Respiratory stability(Able to breathe deeply,Tachypnea,Dyspneic),Hemodynamic stability; (Blood pressure(MAP)<15%, Blood pressure 15-30%, Blood pressure>30%, Level of consciousness,(Awake&orientated Arousable with minimal stimulation, Responsive only to tactile stimulation),Oxygen saturation status(Maintains value>90% on room air, Requires supplemental oxygen, Saturation<90% with supplemental oxygen), Postoperative pain assessment(None or mild discomfort, Moderate to severe pain controlled with analgesics, Persistent severe pain), Postoperative emetic symptoms(None or mild nausea w/no active vomiting, Transient vomiting or retching, Persistent moderate to severe nausea&vomiting), Scoring is done as 2,1,0, respectively. A minimal score of 12(with no score<1 in any individual category)would be required for a patient after general anesthesia
Other: SPEEDS criteria — Extremity movement (moves all four) Y/N, Stable vital signs( SBP > 90 and < 180, HR > 50 and < 110) Y/N, Dialogue (oriented person/place) Y/N, Oxygen saturation >90% in roExtremity movement (moves all four) Y/N, Stable vital signs( SBP > 90 and < 180, HR > 50 and < 110) Y/N, Dialogue (oriented person/place) Y/N, Oxygen saturation >90% in room air Y/N, Pain Control (VAS < 4) Y/N, Emesis Control Y/N. A patient must have a response of "yes" to all parameters to progress to phase II recovery

SUMMARY:
122 ASA I-II patients were enrolled into the study. IV propofol, fentanyl and rocuronium were used for the induction and a total intravenous anesthesia technique for the maintenance of anesthesia. Sugammadex was given for neuromuscular blockade reversal. A multi-modal analgesic regimen was utilized. Primary outcome measures were PACU bypass rates and hospital discharge times. Secondary outcome measure was to compare discharge scoring systems for PACU bypass assessment: modified Aldrete Scoring System (mASS), White's Fast-Tracking Scoring System (WFTSS), and SPEEDS criteria

DETAILED DESCRIPTION:
After obtaining hospital's ethics committee approval (University of Medical Sciences, Gülhane Training and Research Hospital- Date: 06/05/2018; No: 18/148) and written informed consents obtained from patients, 122 ASA (American Society of Anesthesiologists) physical status I-II patients, aged between 18-65 years, undergoing elective lumbar discectomy under general anesthesia were included into the study . After anesthesia application applied to all groups with the same procedure, patients were extubated after surgery. After extubation, patients were evaluated using mASS, WFTSS and SPEEDS criteria during 15 minutes with 3 min intervals. Patients who fulfilled criteria of all scoring systems were defined as eligible for PACU by-pass (fast-tracking) and transferred into phase II recovery area in the ward without observation in PACU (Group FT = Fast Track;). Ineligible patients were taken into PACU where their treatments were continued until discharge criteria were achieved (Group PACU). All patients were followed in the ward until hospital discharge. IV tramadol PCA (Patient -Controlled Analgesia; infusion rate: 4 mgh-1, bolus dose: 4mg, lock-out time: 30 min., 4 hours-limit: 30 mg), paracetamol (10 mgkg-1 IV with 6 hrs. intervals) and oral diclofenac sodium (75 mg with 8 hrs. intervals) were given in a multimodal analgesic regimen. Pain was evaluated using Visual Analogue Scale (VAS) with 2 hours intervals and IV pethidine 0.5 mgkg-1 was given as rescue analgesic throughout the study period when VAS was >3. PONV was treated using IV 4 mg ondansetron. Discharge from hospital was evaluated using Post Anesthetic Discharge Scoring System (PADSS), . Patients with a PADSS score ≥ 9 were discharged from the hospital by the escort of their relatives.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) physical status I-II patients
* elective primary lumbar discectomy performed for one or two vertebra levels under general anesthesia
* minimal risks for perioperative bleeding and airway safety

Exclusion Criteria:

* patient's refusal
* urgent surgery,
* regional anesthesia,
* history of previous lumbar surgery
* difficult ventilation and intubation,
* treatment for chronic pain
* obstructive sleep apnea,
* morbid obesity (BMI≥40 kg/m2)
* allergy to drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 122 ASA (American Society of Anesthesiologists) physical status I-II patients, aged between 18-65 years, undergoing elective lumbar discectomy under general anesthesia were included into the study.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Duration of the surgery | at the end of the surgery
  the period (minutes) from the beginning of the surgery to the end of surgery
time to extubation | 1 hour after extubation
  the period (minutes) from the end of surgery until extubation
PACU( post-anesthesia care unit) by-pass rate | 1 weeks after discharge from the hospital
  The period (minutes) from admission to post-anesthesia care unit to discharge from the clinic
Time to hospital discharge | 1 weeks after discharge from the hospital
  The period (hours) from hospital admission to hospital discharge.
Time to PACU by-pass in group FT | 1 weeks after discharge from the hospital
  time(minutes) to be eligible for PACU by-pass in group FT according to scoring systems
time to PACU care in group PACU | 1 weeks after discharge from the hospital
  duration (minutes) of PACU care for patients in group PACU
patients who were eligible for fast-tracking | through study completion, an average of 2 weeks
  number patients who were eligible for fast-tracking
patients who were discharged from hospital | through study completion, an average of 2 weeks
  number patients who were discharged from hospital with respect to outpatient surgery (discharge time < 24 hours)
factors preventing | through study completion, an average of 2 weeks
  factors preventing fast-tracking and/or discharge from hospital in outpatient setting

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Ö ÖZHAN, M.D., Study Director — Çankaya Hospital, Department of Anesthesiology and Reanimation, Ankara, Turkey; Mehmet B. EŞKİN, M.D., Principal Investigator — Gulhane Training and Research Hospital
Locations (1):
- Çankaya Hospital, Department of Anesthesiology and Reanimation, Ankara, Turkey, Ankara, Çankaya/ANKARA, Turkey (Türkiye)